CLINICAL TRIAL: NCT04107714
Title: Starting the Conversation (STC) - Web-based Group Intervention to Support Disclosure Decisions for Parents of Children With Mental Illness
Brief Title: Starting the Conversation
Acronym: STC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to a small number of study participants.
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Nicolas Rüsch, Professor, University of Ulm
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 375/18
Record Dates: First submitted 2019-09-25; First posted 2019-09-27 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Stigma of Parents of Children With Mental Illness
Keywords: Stigma; Parents of children with mental illness; Disclosure; Secrecy; Group intervention
MeSH Terms: conditions — Social Stigma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (STC) (Experimental): Study participants randomized to the experimental group receive the intervention (STC). STC is a peer-led and web-based group intervention containing four two-hour sessions within four weeks plus an additional booster session one month later.
  Fidelity to manual is rated in each session by study staff.
  Interventions: Behavioral: STC
- No intervention (No Intervention): Participants randomized to the control group do not receive the group program but get the accompanying workbook at the end of the study.

INTERVENTIONS:
Behavioral: STC — The peer-led and web-based group program contains four lessons plus one booster session:
  * Lesson 1: Consider the pros and cons of disclosing: Participants reflect on their experience of self-stigma and weight their pros and cons of (non-)disclosing their child's mental illness.
  * Lesson 2: Different ways to disclose: Participants learn about different ways to disclose and their respective pros and cons. Afterwards participants discuss possible responses they might experience and develop strategies to cope with.
  * Lesson 3: Communication about disclosure between parents and their child: Participants discuss pros and cons of (non-)disclosure for their children and how to negotiate whether to disclose or not.
  * Lesson 4: Telling your story: Participants learn how to tell their own story.
  * In a booster session, participants discuss their experiences with disclosure or non-disclosure.
  Arms: Intervention (STC)

SUMMARY:
The purpose of the study is to evaluate the group-based intervention "Starting the Conversation" as a webinar in Germany. Feasibility and efficacy of the program will be tested in a pilot randomized-controlled trial (RCT).

DETAILED DESCRIPTION:
Parents of children with mental illness often experience public and self-stigma, and keeping a child's mental illness secret is a common strategy to avoid stigma. Both secrecy and disclosure have pros and cons for parents and their children. Therefore, the decision whether, when, and to whom to disclose a child's mental illness is complex. Interventions can provide guidance for systematic consideration and a well informed decision.

The manualized peer-led group intervention "Honest, Open, Proud" (HOP) supports people with mental illness in their decision whether to disclose mental illness. Research showed positive effects of the intervention on stigma stress, disclosure-related distress and quality of life. Based on HOP, "Starting the Conversation" (STC) was developed to systematically guide parents through their decision whether and how to disclose a child's mental illness.

At the moment, there is no data regarding feasibility and efficacy of STC, but two pilot RCTs of STC are currently underway, one in Western Australia and one in Wisconsin, USA. The aim of the current study is to evaluate feasibility and efficacy of STC as a webinar in a pilot RCT in German.

ELIGIBILITY:
Inclusion Criteria:

* Parent with at least one child or adolescent that (i) is aged between 6 to 17 years (ii) has a current mental disorder according to ICD-10 diagnosed by a psychiatrist or psychologist
* Age ≥ 18 years
* Positive screening for disclosure distress (1 item: "In general, how distressed or worried are you in terms of secrecy or disclosure of the mental illness of your child?", self-report, persons with a score ≥ 4 on a scale from 1-7 were included)
* Online informed consent
* Sufficient German language skills

Exclusion Criteria:

* Intellectual disability of child (IQ<70, self-report)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Self-stigma of parents | 8 weeks
  Parent's Self-Stigma Scale (PSSS) (Eaton et al., 2018), 11 items rated from 1 to 5, sum score (range 5-55) with higher scores indicating more self-stigma.

SECONDARY OUTCOMES:
Self-stigma of parents | baseline, 4 weeks, 16 weeks
  Parent's Self-Stigma Scale (PSSS) (Eaton et al., 2018), 11 items rated from 1 to 5, sum score (range 5-55) with higher scores indicating more self-stigma.
Self-stigma of parents | baseline, 4 weeks, 8 weeks, 16 weeks
  Self-Stigma in Relatives of People with Mental Illness Scale (SSRMI) (Morris et al., 2018), 10 items rated from 1 to 5, mean score across all items (range 1-5) with higher scores indicating more self-stigma.
Stigma stress related to child's mental illness | baseline, 4 weeks, 8 weeks, 16 weeks
  Stigma Stress Scale (Rüsch et al., 2009a,b) adapted for parents of children with mental illness, 8 items rated from 1 to 7 with 4 items measuring the primary appraisal of stigma as harmful and 4 items measuring the secondary appraisal of perceived resources to cope with stigma-related harm, for each of the two subscales there is a mean score (range 1-7), and a total stigma stress score will be calculated by subtracting perceived resources from perceived harm with higher difference scores (range -6 to +6) indicating more stigma stress.
Parenting distress | baseline, 4 weeks, 8 weeks, 16 weeks
  Parenting Stress Index, parent domain (PSI) (Tröster, 2011), 28 items rated from 1 to 5, sum scores of subscales (range 4-20) and across all items (range 28-140) with higher scores indicating more parenting distress.
Quality of life of parents | baseline, 4 weeks, 8 weeks, 16 weeks
  World Health Organization Quality of Life Assessment-short form (WHOQOL-BREF), domains general quality of life, psychological and social relationships (Angermeyer, Kilian & Matschinger, 2000), 11 items rated from 1 to 5, mean scores of each domain (range 1-5) with higher scores indicating better quality of life.
Parent-rated child quality of life | baseline, 4 weeks, 8 weeks, 16 weeks
  KIDSCREEN-10, parent version (The KIDSCREEN Group Europe, 2006), 10 items rated from 1 to 5, sum score across all items (range 5-50) with higher scores indicating better child quality of life.
Self-esteem | baseline, 4 weeks, 8 weeks, 16 weeks
  Rosenberg Self-Esteem Scale (RSE) (Collani & Herzberg, 2003), 10 items rated from 0 to 3, sum score across all items (range 0-30) with higher scores indicating higher self-esteem.
Social support | baseline, 4 weeks, 8 weeks, 16 weeks
  Perceived Social Support Questionnaire (FsozU K-6) (Kliem et al., 2015), 6 items rated from 1 to 5, mean score across all items (range 1-5) with higher scores indicating more perceived social support.
Social inclusion | baseline, 4 weeks, 8 weeks, 16 weeks
  Social Inclusion Scale (SIS) (Hacking et al., 2008; Secker et al., 2009) adapted for parents of children with mental illness, 20 items rated from 1 to 4, mean scores (range 1-4) of subscales and across all items with higher scores indicating higher social inclusion.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Child and Adolescent Psychiatry, University of Ulm, Ulm, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eaton K, Ohan JL, Stritzke WGK, Corrigan PW. The Parents' Self-Stigma Scale: Development, Factor Analysis, Reliability, and Validity. Child Psychiatry Hum Dev. 2019 Feb;50(1):83-94. doi: 10.1007/s10578-018-0822-8. PMID 29956016
- [Background] Morris E, Hippman C, Murray G, Michalak EE, Boyd JE, Livingston J, Inglis A, Carrion P, Austin J. Self-Stigma in Relatives of people with Mental Illness scale: development and validation. Br J Psychiatry. 2018 Mar;212(3):169-174. doi: 10.1192/bjp.2017.23. Epub 2018 Feb 5. PMID 29436312
- [Background] Rusch N, Corrigan PW, Powell K, Rajah A, Olschewski M, Wilkniss S, Batia K. A stress-coping model of mental illness stigma: II. Emotional stress responses, coping behavior and outcome. Schizophr Res. 2009 May;110(1-3):65-71. doi: 10.1016/j.schres.2009.01.005. Epub 2009 Feb 23. PMID 19237266
- [Background] Rusch N, Corrigan PW, Wassel A, Michaels P, Olschewski M, Wilkniss S, Batia K. A stress-coping model of mental illness stigma: I. Predictors of cognitive stress appraisal. Schizophr Res. 2009 May;110(1-3):59-64. doi: 10.1016/j.schres.2009.01.006. Epub 2009 Mar 6. PMID 19269140
- [Background] Tröster H. Eltern-Belastungs-Inventar: Deutsche Version des Parenting Stress Index (PSI) von R. R. Abidin [German version of Parenting Stress Index of R. R. Abidin]. Göttingen: Hogrefe; 2011.
- [Background] Angermeyer MC, Kilian R, Matschinger H. WHOQOL-100 und WHOQOL-BREF: Handbuch für die deutschsprachigen Versionen der WHO Instrumente zur Erfassung von Lebensqualität [WHOQOL-100 and WHOQOL-BREF: Handbook for the German version of WHO instruments to assess quality of life]. Göttingen: Hogrefe; 2000.
- [Background] The KIDSCREEN Group Europe. The Kidscreen questionnaires: Quality of life questionnaires for children and adolescents: handbook. Lengerich: Pabst Science Publishers; 2006.
- [Background] Kliem S, Mossle T, Rehbein F, Hellmann DF, Zenger M, Brahler E. A brief form of the Perceived Social Support Questionnaire (F-SozU) was developed, validated, and standardized. J Clin Epidemiol. 2015 May;68(5):551-62. doi: 10.1016/j.jclinepi.2014.11.003. Epub 2014 Nov 13. PMID 25499982
- [Background] Hacking S, Secker J, Spandler H, Kent L, Shenton J. Evaluating the impact of participatory art projects for people with mental health needs. Health Soc Care Community. 2008 Dec;16(6):638-48. doi: 10.1111/j.1365-2524.2008.00789.x. Epub 2008 May 13. PMID 18484974
- [Background] Secker J, Hacking S, Kent L, Shenton J, Spandler H. Development of a measure of social inclusion for arts and mental health project participants. Journal of Mental Health. 2009;18(1):65-72. doi:10.1080/09638230701677803